CLINICAL TRIAL: NCT05116657
Title: Obstructive Sleep Apnoea Post Covid 19: Role of the Upper Airway Microbiome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 21-031
Record Dates: First submitted 2021-11-10; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Sleepiness; SARS-CoV2 Infection; Fatigue Syndrome, Chronic; Snoring
Keywords: sars-CoV2; microbiome; obstructive sleep apnea
MeSH Terms: conditions — Sleepiness; COVID-19; Fatigue Syndrome, Chronic; Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Nasal Lavage: The nasal lavage will be performed using a spray technique. Using a disposable metered-dose inhaler (100 µl per spray), room temperature saline will be sprayed in one nostril while the other nostril is closed. After 5 sprays, the subject will gently exhale through the lavaged nostril and the fluid will be collected in a specimen cup. The procedure will be repeated a minimum of 8 times and a maximum of 15 times in each nostril. After collection, the sample will be placed on ice and processed within 2 hours.
  * Oral Rinse: Oral samples will be collected using a standardized procedure in accordance with the Manual of Procedures for Human Microbiome Project. Study participants will rinse their mouth (swish/gargle) with 15 mL sterile normal saline for 1 min, and will expectorate the contents of the mouth into a 50 mL centrifuge tube. Sample should be kept cold on ice until processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV2 OSA: Patients will be recruited from both Post-COVID19 and Sleep Clinics run through Beaumont Hospital, Beaumont, Dublin, Ireland. This will allow for the recruitment of patients with and without a history of SARS-CoV-2 infection.
  Interventions: Diagnostic Test: Nasal Lavage and Oral Wash
- Non-SARS-CoV2 OSA: Patients will be recruited from both Post-COVID19 and Sleep Clinics run through Beaumont Hospital, Beaumont, Dublin, Ireland. This will allow for the recruitment of patients with and without a history of SARS-CoV-2 infection.
  Interventions: Diagnostic Test: Nasal Lavage and Oral Wash

INTERVENTIONS:
Diagnostic Test: Nasal Lavage and Oral Wash — * Nasal Lavage: The nasal lavage will be performed using a spray technique. Using a disposable metered-dose inhaler (100 µl per spray), room temperature saline will be sprayed in one nostril while the other nostril is closed. After 5 sprays, the subject will gently exhale through the lavaged nostril and the fluid will be collected in a specimen cup. The procedure will be repeated a minimum of 8 times and a maximum of 15 times in each nostril. After collection, the sample will be placed on ice and processed within 2 hours.
  * Oral Rinse: Oral samples will be collected using a standardized procedure in accordance with the Manual of Procedures for Human Microbiome Project.Study participants will rinse their mouth (swish/gargle) with 15 mL sterile normal saline for 1 min, and will expectorate the contents of the mouth into a 50 mL centrifuge tube. Sample should be kept cold on ice until processing.
  Other Names: Home Sleep Study; Positive Airway Pressure if diagnosed with Sleep Apnea

SUMMARY:
Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) causing coronavirus disease, Covid-19, has spread rapidly across the globe since its emergence in January 2020. As of January 2021, there are 87.6 million confirmed cases worldwide, with 1.9milion deaths. In conjunction with this high disease incidence, there have also been reports of Covid-19 related sleep disordered breathing, with up 18% in a Chinese study and 57% in an Italian study of individuals with Covid-19 reporting sleep disturbance.

Obstructive Sleep Apnea (OSA) is a common, chronic condition due to partial or complete upper airway collapse during sleep. OSA is more common in males & obese individuals, both of which are more adversely affected by SARS-CoV-2 infection. Furthermore, inflammation of the upper airway, or nasal passages leading to congestion could lead to a compromised upper airway during sleep and subsequently, obstructive sleep apnea.

We believe that's SARS -CoV-2 infection, and subsequent Covid-19 will lead to an altered microbiome in the upper airway. This is turn will lead to worsening nasal inflammation and congestion, which could predispose individual with previous Covid-19 disease to OSA.

Additionally, OSA is treated with Continuous Positive Airway Pressure (CPAP) a machine which delivers pressurized air into the upper airway via a face mask. This keeps the upper airway open during sleep. When CPAP is well tolerated by individuals, it works well to reduce the symptoms of OSA. Unfortunately, many patients find it difficult to tolerate CPAP. One reason often reported for poor tolerance is nasal congestion. We believe that an altered upper airway microbiome, due to previous SARS-CoV-2 infection, will affect treatment adherence to CPAP therapy. Secondly, we will investigate if treatment with CPAP therapy causes any change in the upper airway microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of sleepiness, fatigue, loud snoring

Exclusion Criteria:

1. Gross skeletal alterations affecting the upper airway (eg.micrognathia)
2. Unstable chronic medical conditions known to affect OSA (CHF, stroke) 3.
3. Pregnancy or intent to become pregnant within the period of the protocol
4. Inability to sign informed consent form
5. Habitual snorer or previous diagnosis of OSA.
6. Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the Sleep Clinic and Post-Covid Clinic in Beaumont Hospital. Participants with snoring and daytime somnolence requiring sleep assessment as part of routine clinical care will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-22 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Examine the incidence of post SARS-CoV-2 infection obstructive sleep apnoea (OSA) and its relationships with the upper airway/nasal microenvironment | 1 year

SECONDARY OUTCOMES:
Determine the relationship between post- SARS-CoV-2 Infection OSA, Positive Airway Pressure (PAP) treatment adherence and change in the upper airway/nasal microenvironment. | 1 year

IPD SHARING:
Plan to Share IPD: No